CLINICAL TRIAL: NCT07040345
Title: Clinical Trial for the Evaluation of Annurca Apple Peel Oleolite for the Treatment of Skin Hyperpigmentation
Brief Title: Annurca Apple Peel Oleolite for the Treatment of Skin Hyperpigmentation
Acronym: EAAO22G01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ritamaria Di Lorenzo (Other)
Responsible Party: Sponsor-Investigator, Ritamaria Di Lorenzo, Principal Investigator, Federico II University
Organization: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EAAO22G01; EAAO22G01 (Other: Institutional Review Board Department of Pharmacy - University of Naples Federico II)
Record Dates: First submitted 2025-06-05; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2023-01

CONDITIONS: Hyperpigmentation; Melasma; Skin Spots; Photodamaged Skin
Keywords: hyperpigmentation; melanogenesis; melasma; skin spots; photodamage
MeSH Terms: conditions — Hyperpigmentation; Melanosis; Exanthema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAO (Active Comparator): Annurca apple oleolite at 2.5% w/w in a cosmetic w/o emulsion twice per day for 28 days
  Interventions: Other: Annurca apple oleolite
- Placebo (Placebo Comparator): cosmetic w/o emulsion without the active comparator twice daily for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Annurca apple oleolite — 3 mg twice daily for 28 days
  Arms: AAO
Other: Placebo — 3 mg twice daily for 28 days
  Arms: Placebo

SUMMARY:
The aim of this cosmetic clinical trial is to learn if an oleolite derived from Annurca Apple peel (AAO) works to enhance skin tone and luminosity, by counteracting the visibility of skin hyperpigmentation and dark spots in adult women with photo-damage. It will also learn about the safety and tolerability of the cosmetic active ingredient. The main questions it aims to answer are:

Does cosmetic active ingredient improve skin tone, luminosity and reduce skin spots visibility? What skin benefits do participants have when using this new active ingredient in a cosmetic formulation? Researchers will compare the AAO to a placebo (a look-alike cosmetic formulation that contains no AAO) to see if AAO works as a depigmenting and whitening ingredient for skin wellness.

Participants will:

Take AAO or a placebo every day twice daily for 28 days (4 weeks) Visit the clinic once every 2 weeks for check-ups and skin parameters observation Keep a diary of the potential adverse reactions that might result from using the assigned test products

DETAILED DESCRIPTION:
The skin effects of the AAO were evaluated through a monocentric, double-blind, placebo-controlled, parallel-arm, randomized clinical study. Healthy Italian subjects (age 40-65; n=48) were enrolled in this 4-week study. Before participating, each subject signed a written informed consent that contained the aim and the type of the study, the list of the cosmetic-grade ingredient employed fort the preparation of the cosmetic formulation, the rules to be followed, and any known or potential adverse reactions that might result from using the test products.

All subjects were selected based on the presence of photodamage and hyperpigmentation. Enrolled subjects underwent to 30-day washout period, in which they were instructed to stop using their usual cosmetic products, whereas they were permitted to continue their normal facial treatment regimen (e.g., facial cleanser, make-up and make-up removal) that did not contain ingredients with lightening or whitening action. Once the wash-out period elapsed, subjects were supplied with test products (placebo and the same formulation added with AAO).

Panelists had to apply the assigned emulsion twice daily (morning and evening) for 4 weeks. The application amount had to be approximately 0.3 g of product (two pumps) on a dry or slightly moistened face. Massage in, avoiding direct contact with the eyes. Upon application, in case of individual hypersensitivity, discontinue treatment. Do not use on irritated or chapped skin. For the evening application wait for at least 1 h before bedtime.

Digital images of all subjects were captured at baseline and at weeks 2 and 4, with VISIA® 7th (Canfield Scientific Inc., Parsippany, NJ 07054 USA). The skin imaging system exploits RGB technology to record and measure UV and brown spots, and skin tone. Before image capture, subjects were equilibrated in a controlled temperature room (22 ± 2 °C) for 30 minutes. The hair of the participants was tied up and their clothing was covered with black cloth. The images were taken by the same operator using the same imaging equipment under the same conditions (lighting, distance, head position, etc.) at all time points. Accurate subjects' repositioning was obtained by comparing the live image with the ghost-baseline digitally stored photo. Computer analysis of the digital images allowed quantification of the hyperpigmentation and dark spots.

Facial skin color and spots were also detected through reflectance and spectro-photometric skin devices, like Skin-Colorimeter® CL 400 and Mexameter® MX 18 (Courage+Khazaka electronic GmbH). Specifically, the skin luminosity, melanin index and skin complexion were monitored during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian subjects
* Age: 18 - 70 years
* Sex: feminine
* Normal adult skin, with spots extinct and wrinkles
* Sensitive skin, with brown spots
* Phototype: II - III Fitzpatrick scale
* Subjects who have read and signed the informed consent written by the investigators
* Subjects who did not apply on the test area other products than the one studied and no product within seven days before the test
* Subjects who have agreed to follow the study rules and the planned check-ups
* Subjects who have agreed not to expose themselves to UV for the study duration

Exclusion Criteria:

* - Pregnant or breastfeeding women
* Subjects with anamnesis of cutaneous hyper-reactivity or intolerance reactions to cosmetic products/ingredients
* Subjects with diseases in the period immediately preceding the current study
* Subjects undergoing topical or systemic treatment with any drug that may affect the outcome of the test or affected by skin diseases (eczema, psoriasis, lesions)
* Subjects receiving topical or oral retinoic acid or any derivative of vitamin A (tretinoin or isotretinoin) in the six months before the start of the study and systemically in the previous 12 months
* Subjects who performed treatments with topical products based on alpha and beta-hydroxy acids, or other whitening agents, the 45 days before the test start
* Subjects who took systemic antiaging and antioxidant supplements within 60 days before the start of the study
* With thyroid disorders (hyperthyroidism/hypothyroidism) and who are not undertaking due treatment, or those taking the medications for less than one year
* Who has received a facial filling in the last 12 months
* Who is doing any facial aesthetic procedure
* Who are using cosmetics or medications that may increase the photosensitivity of the skin
* Who have undergone bariatric surgery or who are confined to a strict diet
* Who is using any supplement (topic or oral) for the improvement of their skin condition

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Depigmenting activity | 28 days
  i) skin tone with Individual Typology Angle (ITA°) ii) hyperpigmentation through Melanin index (A.U.) iii) UV and Brown spots (score) were monitored using Mexameter MX18 after 14 and 28 days of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Napoli, Italy 80131, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No